CLINICAL TRIAL: NCT03565705
Title: Impact of Spinal Anesthesia on Peri-operative Opioid Consumption in Open Abdominal Prostatectomy- a Retrospective Analysis
Brief Title: Spinal Anesthesia and Peri-operative Opioid Consumption in Open Abdominal Prostatectomy
Acronym: SAPOC
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 042017
Record Dates: First submitted 2018-04-24; First posted 2018-06-21 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Pain, Postoperative; Opioid Use; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spinal anesthesia with propofol sedation: Patients receive spinal anesthesia for analgesia to undergo open abdominal prostatectomy. Ventilation is secured via a laryngeal mask under propofol sedation and no muscular blocking is necessary.
  Interventions: Procedure: Open abdominal prostatectomy
- General anesthesia: General anesthesia is conducted with a combination of intravenous opioid (sufentanil) and neuromuscular blocking agent for open abdominal prostatectomy. Patients receive an induction bolus of propofol, undergo tracheal intubation and maintenance of sedation by sevoflurane.
  Interventions: Procedure: Open abdominal prostatectomy

INTERVENTIONS:
Procedure: Open abdominal prostatectomy — Patients undergo standardized open abdominal prostatectomy.

SUMMARY:
Retrospective analysis to assess the impact of spinal anesthesia on peri-operative opioid consumption during open abdominal prostatectomy. The authors compare the group that had spinal anesthesia in combination with propofol sedation and a laryngeal mask to the second group that underwent the same procedure in general anesthesia with tracheal intubation.

DETAILED DESCRIPTION:
Retrospective analysis to assess the impact of spinal anesthesia on peri-operative opioid consumption during open abdominal prostatectomy. The authors compare the group that had spinal anesthesia in combination with propofol sedation and a laryngeal mask to the second group that underwent the same procedure in general anesthesia with tracheal intubation.

...

ELIGIBILITY:
Inclusion Criteria:

* elective, radical abdominal prostatectomy
* >18 years

Exclusion Criteria:

* chronic pain therapy (e.g. out-of-hospital opioid therapy)
* laparoscopic approach

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to include patients that are scheduled for elective, radical open abdominal prostatectomy. Thus only male patients of 18 years or older will participate. Patients with chronic pain therapy (e.g. out-of-hospital opioid therapy) will be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 636 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-10-14 (Actual)

PRIMARY OUTCOMES:
Post-operative opioid consumption | 1 day
  Consumption of piritramid [mg] in PACU.

SECONDARY OUTCOMES:
Intra-operative opioid consumption | 1 day
  Consumption of sufentanil [mg] during surgery. Piritramid is given if NRS score is > 3.
Pain maximum | 1 day
  Postoperative pain level measured with the highest score in numeric pain rating scale (NRS)
Postoperative recovery time | 1 day
  Time interval between postoperative tracheal extubation and the patient reaching fit-for-discharge criteria from the PACU to the ward.
PONV/Shivering | 1 day
  Occurence of post-operative nausea and vomiting or shivering in PACU.

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Nitzschke, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Department of Anesthesiology; Center of Anesthesiology and Intensive Care Medicine, Hamburg Eppendorf University Medical Center, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Funcke S, Schick-Bengardt X, Pinnschmidt HO, Beyer B, Fischer M, Kahl U, Nitzschke R. The impact of spinal anaesthesia on perioperative opioid consumption, postoperative pain and oncological outcome in radical retropubic prostatectomy-a retrospective before-and-after effectiveness study. Perioper Med (Lond). 2022 Oct 3;11(1):49. doi: 10.1186/s13741-022-00281-0. PMID 36184629